CLINICAL TRIAL: NCT07065084
Title: The Effect of Virtual Reality Application on Pain, Anxiety and Vital Signs During the Procedure in Hernia Patients Operated With Spinal Anesthesia
Brief Title: The Effect of Virtual Reality Application on Pain, Anxiety, Vital Signs on Hernia Patients Operated With Spinal Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Celal Bayar University (Other)
Responsible Party: Principal Investigator, Dilek Çeçen Çamlı, Asist. Prof. Dr, Celal Bayar University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 24/11/2021/20.478.486/997
Record Dates: First submitted 2025-04-28; First posted 2025-07-15 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-05

CONDITIONS: Patient Centered Care
Keywords: virtual reality; ağrı; anxiety
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: intervention: one group was shown a video with virtual reality goggles during the surgical intervention.
  control: this group underwent a routine surgical procedure throughout the surgical intervention. No intervention was performed.
  The difference in pain, vital signs and anxiety between the two groups was analyzed.
Masking Description: No additional masking was applied.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study (video wathced with VR glasses) (Experimental): the patients in the intervention group were fitted with VR goggles by the researcher immediately after the spinal anesthesia was administered by the researcher during the operation in hernia patients who received spinal anesthesia for the study, when the patient was placed on the operating table and given the operating position, just before the surgical incision started. The procedures were performed without interfering with anesthesia and general operating room functioning. When the surgical incision was to be made, videos were started to be watched from the VR glasses simultaneously. During the 20 minute procedure, the licensed product "Relax with Nature" with music background with virtual reality glasses
  Interventions: Procedure: Virtual Reality glasses
- Control (routine surgical procedure) (No Intervention): this group underwent a routine surgical procedure throughout the surgical intervention. No intervention was performed.

INTERVENTIONS:
Procedure: Virtual Reality glasses — In the study, the patients in the intervention group were fitted with VR goggles by the researcher immediately after the spinal anesthesia was administered by the researcher during the operation in hernia patients who received spinal anesthesia for the study, when the patient was placed on the operating table and given the operating position, just before the surgical incision started. The procedures were performed without interfering with anesthesia and general operating room functioning. When the surgical incision was to be made, videos were started to be watched from the VR glasses simultaneously. During the 20 minute procedure, the licensed product "Relax with Nature" with music background with virtual reality glasses (Bobo VR Z4 Binocular Glasses and 5.7 inch 1440x2560 pixel screen resolution display unit, China) was watched with virtual reality application. Patients were shown videos of lakes, forests, waterfalls, rivers and beaches. In the studies, it was stated that these videos
  Arms: Study (video wathced with VR glasses)

SUMMARY:
Abstract The aim of this study was to evaluate the effect of virtual reality application on pain, anxiety and vital signs during the procedure. This randomized controlled study included 110 hernia patients who underwent spinal anesthesia in the General Surgery Operating Room of a hospital in the western region of Turkey. Patients were randomly assigned to the experimental group or the control group. Patients in the experimental group (n=55) were shown virtual reality goggles and a music-enhanced video for 20 minutes during the surgical procedure. Patients in the control group (n=55) received standard nursing care. Patients in both groups were evaluated using VAS, State and Trait Anxiety Inventory, and Life Findings Monitoring Form.

Keywords: Virtual Reality simulation, Anxiety, Surgery, Pain, Nursing Care

ELIGIBILITY:
Inclusion Criteria:

diagnosed with hernia spinal anesthesia used

Exclusion Criteria:

psychiatric/mental illness vision/hearing disability general anesthesia used

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2021-11-24 (Actual); Primary Completion 2021-11-24 (Actual); Study Completion 2023-06-23 (Actual)

PRIMARY OUTCOMES:
pain level | preoperative and intraoperative: Two time
  Patients' pain intensity was assessed intraoperatively and postoperatively using the Numerical Rating Scale (NRS). Scale scores range from 0-10.
  A high score indicates an increase in the patient's pain.

SECONDARY OUTCOMES:
Anxiety Level | preoperative and intraoperative: two times
  Anxiety scores of the patients before and after surgery were determined using the 'State-Trait Anxiety Inventory' prepared by Spielberger et al.
  The total score of the scale ranges between 20-80. A total score above 60 indicates severe anxiety. a high score on the scale in the study indicates that the patient's anxiety during and after the procedure is elevated.

CONTACTS AND LOCATIONS:
Overall Officials: DILEK CECEN CAMLI, Principal Investigator — MCBÜ SAĞLIK BİLİMLERİ FAKÜLTESİ
Locations (1):
- Manisa Celal Bayar University, Manisa, YUNUSEMRE, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Reason for not sharing IPD: There is no plan to share IPD because the study was not designed for secondary data use.

REFERENCES:
- See also: Like population — https://dergipark.org.tr/tr/download/article-file/507070
- See also: like methods — https://www.cambridge.org/core/journals/palliative-and-supportive-care/article/virtual-reality-for-improving-pain-and-painrelated-symptoms-in-patients-with-advanced-stage-colorectal-cancer-a-pilot-trial-to-test-feasibility-and-acceptability/468C87F1BD774B363A070F86AB65993D?utm_campaign=shareaholic&utm_medium=copy_link&utm_source=bookmark
- Available data/document: Clinical Study Report: dilek.cecen@cbu.edu.tr — https://cdn.clinicaltrials.gov/large-docs/02/NCT04069702/ICF_000.pdf